CLINICAL TRIAL: NCT00212264
Title: Conservative Treatment of Postprostatectomy Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Patricia Goode, MD, Principal Investigator, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK60044 (completed)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; therapy; prostatectomy; prostate cancer
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Behavior Therapy; Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavioral Therapy (Experimental): Behavioral Therapy (Pelvic floor muscle training, bladder control strategies)
  Interventions: Behavioral: Behavioral Therapy
- Behavioral Therapy Plus Technologies (Experimental): Behavioral therapy plus technologies (home pelvic floor electrical stimulation and biofeedback)
  Interventions: Behavioral: Behavioral Therapy; Device: Pelvic Floor Electrical Stimulation; Behavioral: Biofeedback
- Placebo Comparator (Placebo Comparator): No treatment control
  Interventions: Other: No Treatment

INTERVENTIONS:
Behavioral: Behavioral Therapy — Pelvic Floor Muscle Exercises and Bladder control strategies
  Arms: Behavioral Therapy; Behavioral Therapy Plus Technologies
Device: Pelvic Floor Electrical Stimulation — Pelvic Floor Electrical Stimulation daily for 8 weeks
  Arms: Behavioral Therapy Plus Technologies
Behavioral: Biofeedback — Pelvic Floor Muscle training via biofeedback
  Arms: Behavioral Therapy Plus Technologies
Other: No Treatment — No treatment
  Arms: Placebo Comparator

SUMMARY:
The primary purpose of this study is to test the effectiveness, impact on quality of life, and durability of non-surgical therapies for incontinence persisting at least one year after surgery. The study is a a prospective, controlled, randomized trial comparing an 8-week, multi-component behavioral training program (pelvic floor muscle exercises, self-monitoring with bladder diaries, regular office visits, bladder control techniques, and fluid management) to the same program with the addition of biofeedback and pelvic muscle electrical stimulation.

DETAILED DESCRIPTION:
The primary purpose of this project is to test the effectiveness, impact on quality of life, and durability of conservative therapies for persistent post-prostatectomy urinary incontinence in a prospective, controlled, randomized trial comparing an 8-week, multi-component behavioral training program (pelvic floor muscle exercises, self-monitoring with bladder diaries, regular office visits, bladder control techniques, and fluid management) to the same program with the addition of biofeedback and pelvic muscle electrical stimulation.

The second purpose of the study is to examine and compare the cost-effectiveness of the 8-week, multi-component behavioral training program to the same program with the addition of biofeedback and pelvic floor electrical stimulation.

Prostate cancer is the most common internal cancer in men in the United States. The most common treatment for early disease is radical prostatectomy, the removal of the prostate gland. The two most common sequelae of prostatectomy are incontinence and erectile dysfunction. The incontinence improves and often resolves in the first year after prostatectomy, but surveys of patients show that 40% of men have incontinence severe enough to require pads 1 and 2 years after their surgery. There are currently no randomized, controlled studies of non-surgical treatments for persistent post-prostatectomy incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Involuntary loss of urine that started immediately after radical prostatectomy and has persisted for at least one year.
2. One-week bladder diary with interpretable data and at least two incontinence episodes

Exclusion Criteria:

1. Any unstable medical condition, particularly decompensated congestive heart failure, history of malignant arrhythmias, or unstable angina
2. Cardiac pacemaker or implanted cardiac defibrillator
3. Current use of anticholinergic agents for detrusor instability
4. Folstein's Mini-Mental State Exam score below 24 (impaired mental status)
5. One-week bladder diary with continual leakage - defined as always being damp or wet or unable to quantitate individual accidents.
6. Poorly controlled diabetes, defined as (glycosylated hemoglobin > 9 within last 3 months).
7. Hematuria on microscopic examination. Enrollment will be permitted after urologic evaluation.
8. Urodynamic evaluation: Post-void residual volume greater than 200 mL

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2003-08; Primary Completion 2008-09 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S Goode, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Goode PS, Burgio KL, Johnson TM 2nd, Clay OJ, Roth DL, Markland AD, Burkhardt JH, Issa MM, Lloyd LK. Behavioral therapy with or without biofeedback and pelvic floor electrical stimulation for persistent postprostatectomy incontinence: a randomized controlled trial. JAMA. 2011 Jan 12;305(2):151-9. doi: 10.1001/jama.2010.1972. PMID 21224456
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Therapy | Behavioral Therapy Plus Technologies | Placebo Comparator
Started | 70 | 70 | 68
Completed | 58 | 54 | 64
Not Completed | 12 | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Therapy | Behavioral Therapy Plus Technologies | Placebo Comparator | Total
Number analyzed (Participants) | 70 | 70 | 68 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.5) | 66.8 (7.0) | 66.9 (7.7) | 66.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 70 | 70 | 68 | 208
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 15 | 16 | 50
  White | 51 | 54 | 50 | 155
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Incontinence Episodes per Week [Mean (Standard Deviation); unit: Incontinence Episodes per Week] | 28.1 (22.0) | 25.6 (26.0) | 24.8 (19.9) | 26.2 (22.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Incontinence Episodes on Bladder Diary
Description: [(Baseline incontinence episodes minus 2-month incontinence episodes)/baseline incontinence episodes] x 100%
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: % change in episodes per week
Arm/Group | Behavioral Therapy | Behavioral Therapy Plus Technologies | Placebo Comparator
Number analyzed (Participants) | 70 | 70 | 68
% change in episodes per week | 55 [44 to 66] | 51 [37 to 65] | 24 [10 to 39]
Statistical Analysis 1: Comparison: Behavioral Therapy vs Behavioral Therapy Plus Technologies vs Placebo Comparator; Test type: Superiority or Other; p = .001, ANOVA

2. Primary Outcome: Percent Change in Incontinence Episodes Per Week on Bladder Diary
Description: [(Baseline incontinence episodes minus 12-month incontinence episodes)/baseline incontinence episodes] x 100%
Time Frame: 1 year
Population: This outcome was to measure treatment durability. The no-treatment control group completed the study after the primary outcome was collected at 2 months. At that time, they were offered treatment for this burdensome condition outside the study. Only the 2 active treatment groups continued in the study for 1 full year.
Measure: Mean (95% Confidence Interval); unit: % change in episodes per week
Arm/Group | Behavioral Therapy | Behavioral Therapy Plus Technologies
Number analyzed (Participants) | 70 | 70
% change in episodes per week | 50 [40 to 61] | 59 [45 to 73]
Statistical Analysis 1: Comparison: Behavioral Therapy vs Behavioral Therapy Plus Technologies; Test type: Superiority or Other; p = .32, t-test, 1 sided; Note that the no-treatment control group completed the study after 2 months and was not included in this analysis of treatment effect durability

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Behavioral Therapy | Behavioral Therapy Plus Technologies | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 0/70 | 2/70 | 0/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Behavioral Therapy (N=70) | Behavioral Therapy Plus Technologies (N=70) | Placebo Comparator (N=68)
Irritation of Hemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No